CLINICAL TRIAL: NCT00093444
Title: A Phase I Dose Escalation Study Of Heat Activated Liposome Delivery Of Doxorubicin And Radiofrequency Ablation Of Primary And Metastatic Tumors Of The Liver
Brief Title: Heat Activated Liposomal Doxorubicin and Radiofrequency Ablation in Treating Patients With Primary or Metastatic Liver Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 040263; 04-C-0263; CELSION-10403101; CDR0000387979; NCT00090805 (obsolete NCT alias)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: advanced adult primary liver cancer; liver metastases; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

INTERVENTIONS:
Drug: lyso-thermosensitive liposomal doxorubicin
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal doxorubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiofrequency ablation uses high-frequency electric current to kill tumor cells. Combining radiofrequency ablation with liposomal doxorubicin may increase the effectiveness of the drug and kill more tumor cells.

PURPOSE: This phase I trial is studying the best dose of liposomal doxorubicin when given with radiofrequency ablation in treating patients with primary or metastatic liver tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of heat activated doxorubicin HCl liposome when combined with radiofrequency ablation in patients with primary or metastatic tumors of the liver.
* Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.

OUTLINE: This is a dose-escalation study of heat activated doxorubicin HCl liposome.

Patients receive doxorubicin HCl liposome IV over 30 minutes. Approximately 15 minutes after the beginning of the doxorubicin HCl liposome infusion, patients undergo radiofrequency ablation with needles inserted into the tumor(s) and heated to the target temperature for approximately 12-60 minutes.

Cohorts of 3-6 patients receive escalating doses of heat activated doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

Patients are followed at 28 days, every 3 months for 1 year, and then every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed tumor of the liver

  * Primary or metastatic disease
  * No more than 4 lesions
  * No single lesion > 7 cm in maximum diameter
* Not a candidate for curative surgical resection due to tumor histology or prior surgery

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Platelet count ≥ 75,000/mm^3
* WBC ≥ 1,500/mm^3
* Hemoglobin ≥ 10 g/dL (transfusions to attain levels ≥ 10g/dL allowed)

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* PT or PTT ≤ 1.5 times control (except for patients receiving anticoagulation therapy for an unrelated medical condition [e.g., atrial fibrillation])

Renal

* Creatinine ≤ 2.5 mg/dL

Cardiovascular

* See Hepatic
* Ejection fraction ≥ 50% by MUGA
* No congestive heart failure
* No myocardial infarction within the past 6 months
* No cerebral vascular accident within the past 6 months
* No life-threatening cardiac arrhythmia

Other

* Weight < 136 kg
* Glucose ≤ 300 mg/dL
* No uncontrolled diabetes
* No known serious uncontrolled reaction (e.g., anaphylaxis) to contrast agents used in this study
* No known allergy to egg or egg products
* No other serious medical illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent interferon
* No live vaccines (for immunosuppressed patients only) during and for 30 days after study treatment

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* More than 3 weeks since prior therapy for liver tumor(s)
* More than 3 weeks since prior systemic therapy for non-life-threatening extrahepatic disease and recovered
* No other concurrent systemic therapy
* No administration of any of the following medications during and for 30 days after study treatment:

  * Cyclosporine
  * Phenobarbital
  * Phenytoin
  * Streptozocin
* No concurrent administration of any of the following medications:

  * Amphotericin B by injection
  * Antithyroid agents for overactive thyroid
  * Azathioprine
  * Chloramphenicol
  * Colchicine
  * Flucytosine
  * Ganciclovir
  * Plicamycin
  * Zidovudine
  * Probenecid
  * Sulfinpyrazone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-09; Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of heat-activated doxorubicin HCL liposome
Pharmacokinetics and pharmacodynamics of heat-activated doxorubicin HCL liposome at 15, 30, 45, 60, 75, and 90 minutes; 2, 3, 4, 6, 24, and 46 hours; and 4 and 8 days following infusion

SECONDARY OUTCOMES:
Effects of ablative therapy on tumor blood flow and tumor vascular density as measured by MRI at 28 days following study completion

CONTACTS AND LOCATIONS:
Overall Officials: Bradford Wood, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States
- Queen Mary Hospital - Hong Kong, Hong Kong, China